CLINICAL TRIAL: NCT03537014
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Site Phase 3 Study of the Efficacy and Safety of Manualized MDMA-Assisted Psychotherapy for the Treatment of Severe Posttraumatic Stress Disorder
Brief Title: A Multi-Site Phase 3 Study of MDMA-Assisted Psychotherapy for PTSD (MAPP1)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lykos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MAPP1
Record Dates: First submitted 2018-05-14; First posted 2018-05-25 (Actual); Results first posted 2021-09-16 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Therapeutics; N-Methyl-3,4-methylenedioxyamphetamine

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, between-group comparison of change in PTSD symptoms
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Use of separate databases for outcome measures and safety data. Assessment made by pool of independent raters. Randomization will be managed via an Interactive Web Randomization System (IWRS) based on a centralized randomization schedule developed by an independent third-party vendor to maintain blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MDMA-assisted therapy (Experimental): Administration of 80 or 120 mg midomafetamine HCl with a supplemental dose 1.5 to 2 hours later of 40 or 60 mg midomafetamine HCl, respectively, in combination with therapy during 3 experimental sessions scheduled 3-5 weeks apart.
  Interventions: Behavioral: Therapy; Drug: midomafetamine HCl
- Placebo with therapy (Placebo Comparator): Administration of inactive placebo in combination with therapy during 3 experimental sessions scheduled 3-5 weeks apart
  Interventions: Behavioral: Therapy; Drug: Placebo

INTERVENTIONS:
Behavioral: Therapy — Non-directive therapy performed by therapist team
  Other Names: Manualized therapy
Drug: midomafetamine HCl — Administration of 80 to 120 mg midomafetamine HCl, followed by a supplemental dose 1.5 to 2 hrs later of 40 or 60 mg midomafetamine HCl, respectively, during three experimental sessions
  Other Names: 3,4-methylenedioxymethamphetamine; MDMA; midomafetamine; MDMA HCl
  Arms: MDMA-assisted therapy
Drug: Placebo — Administration of placebo during three experimental sessions
  Other Names: Inactive placebo
  Arms: Placebo with therapy

SUMMARY:
The goal of this clinical trial is to learn if MDMA-assisted therapy is safe and effective in people with at least severe PTSD.

The main question it aims to answer is: Do three sessions of MDMA-assisted therapy reduce PTSD symptoms?

Researchers will compare three sessions of MDMA-assisted therapy with an initial dose of 80 to 120 mg to three sessions of placebo with therapy.

Participants will undergo three preparatory sessions without any study drug, followed by three MDMA-assisted therapy or placebo with therapy sessions. Each medication session will be followed by three integrative therapy sessions without study drug.

DETAILED DESCRIPTION:
This multi-site, double-blind, placebo-controlled, randomized Phase 3 study will assess the efficacy and safety of MDMA-assisted therapy versus placebo with therapy in participants diagnosed with at least severe PTSD. The study will be conducted in N ≈ 100 participants. Participants will be randomized to one of two groups at a 1:1 ratio. An initial dose of midomafetamine HCl or placebo, followed by a supplemental half-dose unless contraindicated, is administered during the Treatment Period with manualized therapy in three monthly Experimental Sessions. This ~12-week Treatment Period is preceded by three Preparatory Sessions. During the Treatment Period, each Experimental Session is followed by three Integrative Sessions of non-drug psychotherapy. Initial doses per Experimental Session include 80 mg or 120 mg of midomafetamine HCl or placebo followed 1.5 to 2 hours later by a supplemental half-dose (40 or 60 mg). Total amounts of midomafetamine HCl to be administered per Experimental Session range from 80 mg to 180 mg.

The primary endpoint is change from baseline in Clinician Administered PTSD Scale for DSM-V (CAPS-5) to 18 weeks post-Baseline. Drug safety will be assessed by measuring blood pressure, heart rate and body temperature during Experimental Sessions, collecting adverse events and measuring suicidal thoughts or behaviors with the Columbia Suicide Severity Rating Scale (adapted C-SSRS).

ELIGIBILITY:
Inclusion Criteria:

* Are at least 18 years old
* Are fluent in speaking and reading the predominantly used or recognized language of the study site
* Are able to swallow pills
* Agree to have study visits recorded, including Experimental Sessions, Independent Rater assessments, and non-drug psychotherapy sessions
* Must provide a contact (relative, spouse, close friend or other caregiver) who is willing and able to be reached by the investigators in the event of a participant becoming suicidal or unreachable.
* Must agree to inform the investigators within 48 hours of any medical conditions and procedures
* If of childbearing potential, must have a negative pregnancy test at study entry and prior to each Experimental Session, and must agree to use adequate birth control through 10 days after the last Experimental Session.
* Must not participate in any other interventional clinical trials during the duration of the study
* Must be willing to remain overnight at the study site after each Experimental Session and be driven home after, and commit to medication dosing, therapy, and study procedures
* At baseline, meet DSM-5 criteria for current severe PTSD

Exclusion Criteria:

* Are not able to give adequate informed consent
* Have uncontrolled hypertension
* Have a marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 milliseconds [ms] in males and >460 ms in females corrected by Bazett's formula)
* Have a history of additional risk factors for Torsade de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
* Have evidence or history of significant medical disorders, such as myocardial infarction, cerebrovascular accident, or aneurysm
* Have symptomatic liver disease
* Have history of hyponatremia or hyperthermia
* Weigh less than 48 kilograms (kg)
* Are pregnant or nursing, or are of childbearing potential and are not practicing an effective means of birth control
* Have an active illicit or prescription drug use disorder
* Have used Ecstasy (material represented as containing MDMA) more than 10 times within the last 10 years or at least once within 6 months of the first Experimental Session; or have previously participated in a MAPS-sponsored MDMA clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2020-08-11 (Actual); Study Completion 2020-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Casey Paleos, MD, Principal Investigator — Affective Care; Bessel van der Kolk, MD, Principal Investigator — Trauma Research Foundation; Emma Hapke, MD, Principal Investigator — Dr. Simon Amar, Inc.; Revital Amiaz, MD, Principal Investigator — The Chaim Sheba Medical Center, Tel Hashomer Hospital; Michael Bogenschutz, MD, Principal Investigator — New York University/Langone Medical Center/Bellevue Hospital; Randall Brown, MD, PhD, Principal Investigator — University of Wisconsin, Madison; Sylvestre Quevedo, MD, Principal Investigator — San Francisco Insight and Integration Center; Josh Woolley, MD, PhD, Principal Investigator — University of California, San Francisco; Ray Worthy, MD, Principal Investigator — Ray Worthy Psychiatry, LLC; Cole Marta, MD, Principal Investigator — New School Research, LLC; Scott Shannon, MD, Principal Investigator — Wholeness Center; Wael Garas, MD, Principal Investigator — Aguazul-Bluewater, Inc.; Yevgeniy Gelfand, MD, Principal Investigator — Zen Therapeutics Solutions, LLC
Locations (15):
- United States (11):
  - New School Research LLT, North Hollywood, California
  - San Francisco Insight and Integration Center, San Francisco, California
  - University of California San Francisco, San Francisco, California
  - Aguazul-Blue Water Inc., Boulder, Colorado
  - Wholeness Center, Fort Collins, Colorado
  - Ray Worthy Psychiatry LLC, New Orleans, Louisiana
  - Trauma Research Foundation, Boston, Massachusetts
  - New York University, New York, New York
  - New York Private Practice, New York, New York
  - Zen Therapeutic Solutions, LLC, Mt. Pleasant, South Carolina
  - University of Wisconsin at Madison, Madison, Wisconsin
- Canada (2):
  - Providence Health Center, Vancouver, British Columbia
  - Dr. Simon Amar, Inc., Montreal, Quebec
- Israel (2):
  - Assaf Harofeh Research Fund, Be’er Ya‘aqov
  - Sheba Fund for Health Services and Research, Tel Litwinsky

IPD SHARING:
Plan to Share IPD: Yes
We will share outcome data appearing in any published reports upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data and study-related documents will be available when the database has been locked and data has been unblinded.
Access Criteria: Interested persons should correspond with the central contact for the multisite study.

REFERENCES:
- [Result] Mitchell JM, Bogenschutz M, Lilienstein A, Harrison C, Kleiman S, Parker-Guilbert K, Ot'alora G M, Garas W, Paleos C, Gorman I, Nicholas C, Mithoefer M, Carlin S, Poulter B, Mithoefer A, Quevedo S, Wells G, Klaire SS, van der Kolk B, Tzarfaty K, Amiaz R, Worthy R, Shannon S, Woolley JD, Marta C, Gelfand Y, Hapke E, Amar S, Wallach Y, Brown R, Hamilton S, Wang JB, Coker A, Matthews R, de Boer A, Yazar-Klosinski B, Emerson A, Doblin R. MDMA-assisted therapy for severe PTSD: a randomized, double-blind, placebo-controlled phase 3 study. Nat Med. 2021 Jun;27(6):1025-1033. doi: 10.1038/s41591-021-01336-3. Epub 2021 May 10. PMID 33972795

RESULTS

PARTICIPANT FLOW:
Groups:
- MDMA-assisted Therapy: Administration of 80 or 120 mg MDMA in combination with psychotherapy and a supplemental dose offered 1.5/2 hrs later of 40 or 60 mg MDMA respectively.
  Psychotherapy: Standardized non-directive psychotherapy performed by therapist team
  MDMA: Administration of 80 to 120 mg MDMA during three sessions of MDMA-assisted psychotherapy followed by a supplemental dose of 40 or 60 mg MDMA offered 1.5/2 hrs after the initial dose, respectively.
- Placebo With Therapy: Administration of inactive placebo in combination with psychotherapy
  Psychotherapy: Standardized non-directive psychotherapy performed by therapist team
  Placebo: Administration of placebo during three sessions of MDMA-assisted psychotherapy
Period: Overall Study
Arm/Group | MDMA-assisted Therapy | Placebo With Therapy
Started | 46 | 45
Completed (Completed all study visits) | 42 | 37
Not Completed | 4 | 8

BASELINE CHARACTERISTICS:
Population: Safety set
Groups:
- Total: Total of all reporting groups
Arm/Group | MDMA-assisted Therapy | Placebo With Therapy | Total
Number analyzed (Participants) | 46 | 44 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.55 (12.86) | 38.19 (10.36) | 40.93 (11.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 32 | 59
  Male | 19 | 12 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 41 | 40 | 81
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 2 | 5 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 39 | 30 | 69
  More than one race | 2 | 6 | 8
  Unknown or Not Reported | 0 | 1 | 1
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 26.0 (4.8) | 24.8 (4.2) | 25.4 (4.5)
Duration of PTSD [Mean (Standard Deviation); unit: years] | 14.8 (11.6) | 13.3 (11.4) | 14.0 (11.5)
Dissociative subtype of PTSD [Count of Participants; unit: Participants] | 6 | 13 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Primary Endpoint in Clinician Administered PTSD Scale for DSM-V (CAPS-5)
Description: The CAPS-5 is a 30-item semi-structured interview assessing PTSD in the past month through diagnostic and symptom severity scores anchored to a DSM-5 defined traumatic event. The CAPS-5 produces a Total Severity Score based on severity of PTSD domains described in the DSM-5, as well as a categorical rating indicating whether a participant meets PTSD diagnostic criteria. CAPS-5 Total Symptom Severity scores range from 0 to 80 with higher values indicating greater symptom severity. CAPS-5 assigns PTSD diagnosis as being present or absent.
Time Frame: Baseline to 18 weeks post enrollment confirmation
Population: Modified intention-to-treat
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- MDMA-assisted Therapy: Administration of 80 or 120 mg midomafetamine HCl in combination with psychotherapy and a supplemental dose offered 1.5/2 hrs later of 40 or 60 mg respectively.
Arm/Group | MDMA-assisted Therapy | Placebo With Therapy
Number analyzed (Participants) | 46 | 44
score on a scale | -24.5 [-28.28 to -20.71] | -12.64 [-16.61 to -8.66]

2. Secondary Outcome: Change From Baseline to Primary Endpoint in Sheehan Disability Scale (SDS) Total Score
Description: The Sheehan Disability Scale (SDS) is a clinician-rated assessment of functional impairment that was adapted for the purposes of this study to limit missing item-level data as per the FDA requirements and included use of the three-item mean as the total score and imputation of work-related impairment. The SDS is a 3-item scale measuring the severity of disability in the domains of work, family life/home responsibilities and social/leisure activities, with each item scored on a ten-point Likert scale from 0 ('not at all impaired') to 10 ('very severely impaired'). The SDS total score was the mean of the 3 item responses. The SDS total score ranged from 0 to 10, with higher scores indicating greater functional impairment.
Time Frame: Baseline to 18 weeks post enrollment confirmation
Population: Modified intention-to-treat
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | MDMA-assisted Therapy | Placebo With Therapy
Number analyzed (Participants) | 46 | 44
score on a scale | -3.15 [-3.90 to -2.40] | -1.79 [-2.58 to -1.00]

ADVERSE EVENTS:
Time Frame: During the Treatment Period from the first Experimental Session to the Termination visit (approximately 18 weeks)
Groups:
- MDMA-assisted Therapy: Administration of 80 or 120 mg midomafetamine HCl in combination with manualized psychotherapy and a supplemental dose offered 1.5/2 hrs later of 40 or 60 mg respectively.
- Placebo With Therapy: Administration of inactive placebo in combination with manualized psychotherapy
Arm/Group | MDMA-assisted Therapy | Placebo With Therapy
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/46 | 2/44
Other Adverse Events (participants affected / at risk) | 46/46 | 44/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MDMA-assisted Therapy (N=46) | Placebo With Therapy (N=44)
Suicide Attempt (Psychiatric disorders) | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MDMA-assisted Therapy (N=46) | Placebo With Therapy (N=44)
Palpitations (Cardiac disorders) | 4 | 6
Mydriasis (Eye disorders) | 7 | 0
Vision Blurred (Eye disorders) | 4 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 6 | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 5 | 4
Diarrhea (Gastrointestinal disorders) | 2 | 5
Dry Mouth (Gastrointestinal disorders) | 5 | 2
Nausea (Gastrointestinal disorders) | 14 | 5
Vomiting (Gastrointestinal disorders) | 4 | 0
Asthenia (General disorders) | 5 | 3
Chills (General disorders) | 3 | 0
Crying (General disorders) | 0 | 3
Fatigue (General disorders) | 14 | 14
Feeling Cold (General disorders) | 9 | 3
Feeling Hot (General disorders) | 4 | 4
Feeling Jittery (General disorders) | 5 | 0
Influenza Like Illness (General disorders) | 2 | 3
Non-Cardiac Chest Pain (General disorders) | 4 | 1
Pain (General disorders) | 4 | 1
Pyrexia (General disorders) | 3 | 1
Temperature Intolerence (General disorders) | 4 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 5 | 4
Blood Pressure Increased (Investigations) | 5 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 24 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 4
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 28 | 6
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 3 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 3 | 3
Disturbance in Attention (Nervous system disorders) | 4 | 3
Dizziness (Nervous system disorders) | 9 | 5
Dizziness Postural (Nervous system disorders) | 6 | 2
Headache (Nervous system disorders) | 33 | 24
Hypoaesthesia (Nervous system disorders) | 3 | 2
Nystagmus (Nervous system disorders) | 6 | 0
Paraesthesia (Nervous system disorders) | 5 | 3
Somnolence (Nervous system disorders) | 3 | 0
Tremor (Nervous system disorders) | 5 | 3
Agitation (Psychiatric disorders) | 2 | 3
Anger (Psychiatric disorders) | 3 | 6
Anxiety (Psychiatric disorders) | 15 | 17
Bruxism (Psychiatric disorders) | 6 | 1
Depressed Mood (Psychiatric disorders) | 5 | 4
Depression (Psychiatric disorders) | 4 | 4
Emotional Disorder (Psychiatric disorders) | 2 | 4
Flashback (Psychiatric disorders) | 3 | 2
Insomnia (Psychiatric disorders) | 20 | 13
Intentional Self-Injury (Psychiatric disorders) | 1 | 4
Intrusive Thoughts (Psychiatric disorders) | 4 | 0
Irritability (Psychiatric disorders) | 2 | 5
Nervousness (Psychiatric disorders) | 3 | 0
Nightmare (Psychiatric disorders) | 7 | 7
Restlessness (Psychiatric disorders) | 7 | 0
Stress (Psychiatric disorders) | 4 | 0
Suicidal Ideation (Psychiatric disorders) | 21 | 21
Micturition Urgency (Renal and urinary disorders) | 3 | 0
Pollakiuria (Renal and urinary disorders) | 4 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 10 | 1
Substance Use (Social circumstances) | 3 | 0
Nasopharyngitis (Infections and infestations) | 8 | 6
Panic Reaction (Psychiatric disorders) | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-05-22): https://cdn.clinicaltrials.gov/large-docs/14/NCT03537014/Prot_004.pdf
  • Statistical Analysis Plan (2020-05-22): https://cdn.clinicaltrials.gov/large-docs/14/NCT03537014/SAP_002.pdf
  • Informed Consent Form (2020-06-12): https://cdn.clinicaltrials.gov/large-docs/14/NCT03537014/ICF_005.pdf